CLINICAL TRIAL: NCT02591732
Title: A Nation-wide Registry Study of Patients With Non-valvular Atrial Fibrillation Initiating Anticoagulation Therapies in the Early Period Follow Apixaban Marketing in Denmark: Patient Characteristics, Treatment Patterns, and Early Bleeding Events
Brief Title: A Nationwide Registry Study of Patients With Nonvalvular Atrial Fibrillation Initiating Oral Anticoagulation Therapies In The Early Period Following Apixaban Marketing In Denmark
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: CV185-377
Record Dates: First submitted 2015-10-08; First posted 2015-10-30 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient treated with Apixaban
- Patient treated with Rivaroxaban
- Patient treated with Dabigatran
- Patient treated with vitamin K antagonists

SUMMARY:
The purpose of this study is to describe the characteristics of patients treated with different OATs and whether these characteristics differ between treatments.

Furthermore to describe persistence to each OAT and risk of bleeding after initiating each OAT.

ELIGIBILITY:
Inclusion Criteria:

The study population will consist of all patients in Denmark who meet the following criteria:

* Adult (≥18 years) at time of anticoagulant initiation
* Diagnosed with atrial fibrillation without recorded valvular disease
* Initiated a new OAT during the study period (January 1, 2011 and December 31, 2014).
* For the identification of NVAF cases, the appearance at least one hospital discharge diagnosis of AF will be searched in the databases.

Exclusion Criteria:

* Patients with prosthetic heart valves , rheumatic mitral or aortic valve disorders, and mitral aortic stenosis will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject must be over 18 years of age, male and females are eligible
Sampling Method: Non-Probability Sample
Enrollment: 52178 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The sociodemographic characteristics of all patients with nonvalvular atrial fibrillation (NVAF) who initiated an OAT based on data available in Danish National Patient Registry | Approximately 4 years
  Sociodemographic characteristics: Age,sex, ethnicity, region of residence, education, income and employment status
Clinical characteristics of all patients with NVAF who initiated an Oral anticoagulant therapy (OAT) based on data available in Danish National Patient Registry | Approximately 4 years
  Clinical characteristics: Myocardial infarction, Stroke, Thromboembolism, Hypertension, Peripheral artery disease, Congestive cardiac failure
Previous Oral anticoagulant therapy of all patients with NVAF who initiated an OAT based on data available in Danish National Patient Registry | Approximately 4 years
  Oral anticoagulant: Apixaban, Dabigatran, Rivaroxaban and Vitamin K antagonist
Concomitant medications of all patients with NVAF who initiated an OAT based on data available in Danish National Patient Registry | Approximately 4 years
  Concomitant medication Drug classes: Anti-arrhythmic agents, Antidiabetic agents, Antihypertensive agents, Proton pump inhibitors

SECONDARY OUTCOMES:
Persistence to each OAT after initiation as monotherapy | Approximately 4 years
  Persistence will be defined as treatment discontinuation and will be measured by estimating the following:
  Discontinuation - the absence of any delivery of this product and of any other anticoagulation therapy of interest for 30 days. The date of discontinuation the OAT will be determined according to predefined algorithms to calculate treatment duration in the national prescription registry. Sensitivity analysis including a 30 and 60 day grace period will be performed to take into account incomplete adherence to treatment and dose modifications
Persistence between apixaban and other OAT | Approximately 4 years
  Oral anticoagulant: Dabigatran, Rivaroxaban and Vitamin K antagonist
Clinically relevant bleeding events after initiating an OAT as monotherapy | Approximately 4 years
Bleeding events requiring hospitalization in patients treated with apixaban | Approximately 4 years
Bleeding events requiring out-patient care in patients treated with apixaban | Approximately 4 years
Bleeding events requiring hospitalization in patients treated with rivaroxaban | Approximately 4 years
Bleeding events requiring out-patient care in patients treated with rivaroxaban | Approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hellerup, Denmark

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx